CLINICAL TRIAL: NCT05341622
Title: Pragmatic Trial of Behavioral Interventions to Increase Response to Mailed FIT Outreach
Brief Title: Mailed FIT Outreach 2022
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Principal Investigator, Shivan Mehta, Principal Investigator, Abramson Cancer Center at Penn Medicine
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: UPCC 08222
Record Dates: First submitted 2022-04-18; First posted 2022-04-22 (Actual); Results first posted 2024-07-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Colorectal Cancer; Colon Cancer
Keywords: prevention; cancer screening; mailed FIT
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — Communication Devices for People with Disabilities

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Arm 1: Box + Text + Reminder (Experimental): Box + Text + Reminder
  Interventions: Behavioral: Differentiated Box; Behavioral: Text; Behavioral: Reminder
- Arm 2: Box + Text + No Reminder (Experimental): Box + Text + No Reminder
  Interventions: Behavioral: Differentiated Box; Behavioral: Text; Behavioral: No Reminder
- Arm 3: Box + No Text + Reminder (Experimental): Box + No Text + Reminder
  Interventions: Behavioral: Differentiated Box; Behavioral: No Text; Behavioral: Reminder
- Arm 4: Box + No Text + No Reminder (Experimental): Box + No Text + No Reminder
  Interventions: Behavioral: Differentiated Box; Behavioral: No Text; Behavioral: No Reminder
- Arm 5: Standard Mail + Text + Reminder (Experimental): Standard Mail + Text + Reminder
  Interventions: Behavioral: Standard Mail; Behavioral: Text; Behavioral: Reminder
- Arm 6: Standard Mail + Text + No Reminder (Experimental): Standard Mail + Text + No Reminder
  Interventions: Behavioral: Standard Mail; Behavioral: Text; Behavioral: No Reminder
- Arm 7: Standard Mail + No Text + Reminder (Experimental)
  Interventions: Behavioral: Standard Mail; Behavioral: No Text; Behavioral: Reminder
- Arm 8: Standard Mail + No Text + No Reminder (Experimental): Standard Mail + No Text + No Reminder
  Interventions: Behavioral: Standard Mail; Behavioral: No Text; Behavioral: No Reminder

INTERVENTIONS:
Behavioral: Differentiated Box — Patients will receive mailed FIT kits in a box with differentiated packaging
  Arms: Arm 1: Box + Text + Reminder; Arm 2: Box + Text + No Reminder; Arm 3: Box + No Text + Reminder; Arm 4: Box + No Text + No Reminder
Behavioral: Standard Mail — Patients will receive mailed FIT in a standard mailing envelope
  Arms: Arm 5: Standard Mail + Text + Reminder; Arm 6: Standard Mail + Text + No Reminder; Arm 7: Standard Mail + No Text + Reminder; Arm 8: Standard Mail + No Text + No Reminder
Behavioral: Text — Patients will receive a series of up to 3 texts explaining the importance of colon cancer screening and prompts to complete the mailed FIT.
  Arms: Arm 1: Box + Text + Reminder; Arm 2: Box + Text + No Reminder; Arm 5: Standard Mail + Text + Reminder; Arm 6: Standard Mail + Text + No Reminder
Behavioral: No Text — Patients will not receive text messaging explaining the importance of colon cancer screening or prompts to complete the mailed FIT.
  Arms: Arm 3: Box + No Text + Reminder; Arm 4: Box + No Text + No Reminder; Arm 7: Standard Mail + No Text + Reminder; Arm 8: Standard Mail + No Text + No Reminder
Behavioral: Reminder — Patients will receive a mailed letter reminder to complete their FIT kit if not resulted by 1 month from initial outreach.
  Arms: Arm 1: Box + Text + Reminder; Arm 3: Box + No Text + Reminder; Arm 5: Standard Mail + Text + Reminder; Arm 7: Standard Mail + No Text + Reminder
Behavioral: No Reminder — Patients will not receive any mailed letter reminder to complete their FIT kit.
  Arms: Arm 2: Box + Text + No Reminder; Arm 4: Box + No Text + No Reminder; Arm 6: Standard Mail + Text + No Reminder; Arm 8: Standard Mail + No Text + No Reminder

SUMMARY:
This project aims to evaluate different approaches to increase colorectal cancer screening among primary care patients at Penn Medicine through a centralized screening outreach program. In a pragmatic trial, we will evaluate different approaches to increase response rate to mailed fecal immunochemical test (FIT) kits among eligible patients, including differentiated packaging, sending text reminders, and personalized reminders.

DETAILED DESCRIPTION:
While colonoscopy procedures are recommended by guidelines for early detection of colorectal cancer, colonoscopy access remains limited due to delays in screening due to the pandemic and capacity issues. In this project, we will evaluate different ways of reaching out to eligible patients to encourage them to participate in colorectal cancer screening using fecal immunochemical testing (FIT). In a mailed FIT outreach campaign, we will compare user friendly packaging, text messaging, and personalized reminders to standard outreach with the goal of increasing colorectal cancer screening uptake.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ages 50-74 with Penn as preferred lab
2. Followed by Primary Care with a participating Penn Medicine PCP listed and at least one visit in the last 2 years
3. Not up to date on colorectal cancer screening per Health Maintenance (no colonoscopy in the last 10 years, stool testing in the last year, flexible sigmoidoscopy in the last 5 years, FIT-DNA in the last 3 years).

Exclusion Criteria:

1. Personal or significant family history of CRC, colonic polyps, hereditary nonpolyposis colorectal cancer syndrome, familial adenomatous polyposis syndrome, other gastrointestinal cancer, gastrointestinal bleeding, iron-deficiency anemia, or inflammatory bowel disease
2. History of total colectomy, dementia or metastatic cancer
3. Currently on hospice or receiving palliative care
4. Uninsured or self-pay patients
5. Currently scheduled for a colonoscopy or sigmoidoscopy

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5460 (Actual)
Dates: Start 2022-05-27 (Actual); Primary Completion 2022-10-13 (Actual); Study Completion 2022-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shivan Mehta, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Penn Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mehta SJ, Nadella P, Shaw PA, Reitz C, Brophy C, Okorie E, Williams K, Snider CK, Peifer MK, Rhodes C, Asch DA. Behavioral Interventions Improve Mailed Colorectal Cancer Screening Among Overdue Patients in a Randomized Trial. Clin Gastroenterol Hepatol. 2025 Sep 20:S1542-3565(25)00835-3. doi: 10.1016/j.cgh.2025.09.015. Online ahead of print. PMID 40983155

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1: Box + Text + Reminder | Arm 2: Box + Text + No Reminder | Arm 3: Box + No Text + Reminder | Arm 4: Box + No Text + No Reminder | Arm 5: Standard Mail + Text + Reminder | Arm 6: Standard Mail + Text + No Reminder | Arm 7: Standard Mail + No Text + Reminder | Arm 8: Standard Mail + No Text + No Reminder
Started | 682 | 683 | 681 | 685 | 685 | 687 | 681 | 676
Completed | 656 | 661 | 653 | 661 | 655 | 656 | 653 | 649
Not Completed | 26 | 22 | 28 | 24 | 30 | 31 | 28 | 27
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Invalid Address | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Ineligible | 26 | 21 | 28 | 24 | 29 | 31 | 28 | 26

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Box + Text + Reminder | Arm 2: Box + Text + No Reminder | Arm 3: Box + No Text + Reminder | Arm 4: Box + No Text + No Reminder | Arm 5: Standard Mail + Text + Reminder | Arm 6: Standard Mail + Text + No Reminder | Arm 7: Standard Mail + No Text + Reminder | Arm 8: Standard Mail + No Text + No Reminder | Total
Number analyzed (Participants) | 656 | 661 | 653 | 661 | 655 | 656 | 653 | 649 | 5244
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (7.2) | 60.0 (7.4) | 59.7 (7.4) | 59.6 (7.5) | 59.8 (7.3) | 59.1 (7.1) | 59.9 (7.3) | 59.5 (7.2) | 59.6 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 376 | 377 | 391 | 388 | 366 | 352 | 375 | 371 | 2996
  Male | 280 | 284 | 262 | 273 | 289 | 304 | 278 | 278 | 2248
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 30 | 21 | 32 | 32 | 28 | 27 | 15 | 208
  Not Hispanic or Latino | 619 | 620 | 619 | 616 | 601 | 619 | 616 | 615 | 4925
  Unknown or Not Reported | 14 | 11 | 13 | 13 | 22 | 9 | 10 | 19 | 111
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 3 | 3 | 2 | 0 | 4 | 4 | 3 | 21
  Asian | 30 | 27 | 35 | 22 | 29 | 26 | 26 | 25 | 220
  Native Hawaiian or Other Pacific Islander | 2 | 3 | 1 | 1 | 2 | 0 | 2 | 4 | 15
  Black or African American | 226 | 221 | 241 | 242 | 239 | 238 | 242 | 229 | 1878
  White | 357 | 369 | 342 | 342 | 345 | 332 | 349 | 344 | 2780
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 39 | 38 | 31 | 52 | 40 | 56 | 30 | 44 | 330
Patient Portal Status [Count of Participants; unit: Participants]
  Active | 549 | 555 | 544 | 557 | 553 | 556 | 555 | 542 | 4411
  Not Active | 107 | 106 | 109 | 104 | 102 | 100 | 98 | 107 | 833
Prior Screening (Any) [Count of Participants; unit: Participants] | 188 | 195 | 212 | 192 | 194 | 187 | 210 | 178 | 1556
Insurance Type [Count of Participants; unit: Participants]
  Commercial | 388 | 371 | 392 | 369 | 369 | 371 | 360 | 373 | 2993
  Medicare | 175 | 208 | 172 | 197 | 191 | 186 | 185 | 177 | 1491
  Medicaid | 77 | 71 | 73 | 80 | 84 | 84 | 91 | 84 | 644
  Unknown | 16 | 11 | 16 | 15 | 11 | 15 | 17 | 15 | 116
Median Household Income [Median (Inter-Quartile Range); unit: dollars] | 76973 [39672 to 104232] | 77091 [46698 to 104232] | 77091 [46698 to 104232] | 76854 [39672 to 104232] | 74349 [39672 to 104232] | 77091 [39672 to 104232] | 76610 [43556 to 104232] | 73762 [39672 to 104232] | 76875 [41523 to 104232]

OUTCOME MEASURES:

1. Primary Outcome: FIT Completion
Description: Percent of patients who complete FIT
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Groups:
- Box (Arms 1+2+3+4): All patients in this study arm received mailed FIT in a stylized box. This combined study arm combines all patients in Arms 1-4.
- Envelope (Arms 5+6+7+8): All patients in this study arm received mailed FIT in a plain mailing envelope. This combined study arm includes all patients in arms 5, 6, 7, and 8)
- Text (Arms 1+2+5+6): All patients in this study arm received text messaging related to completion of mailed FIT. This combined study arm includes all patients in study arms 1, 2, 5, and 6).
- No Text (Arms 3+4+7+8): Patients in this study arm did NOT receive any text messaging related to completion of mailed FIT. This combined study arm includes all patients in study arms 3, 4, 7, and 8).
- Reminder (Arms 1+3+5+7): Patients in this study arm did received a mailed reminder letter related to completion of mailed FIT. This combined study arm includes all patients in study arms 1, 3, 5, and 7.
- No Reminder (Arms 2+4+6+8): Patients in this study arm did NOT receive any mailed reminder letters related to completion of mailed FIT. This combined study arm includes all patients in study arms 2, 4, 6, and 8.
Arm/Group | Box (Arms 1+2+3+4) | Envelope (Arms 5+6+7+8) | Text (Arms 1+2+5+6) | No Text (Arms 3+4+7+8) | Reminder (Arms 1+3+5+7) | No Reminder (Arms 2+4+6+8)
Number analyzed (Participants) | 2631 | 2613 | 2628 | 2616 | 2617 | 2627
Participants | 469 | 470 | 558 | 381 | 532 | 407

2. Secondary Outcome: FIT Completion
Description: Percent of patients who complete FIT
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Box (Arms 1+2+3+4) | Envelope (Arms 5+6+7+8) | Text (Arms 1+2+5+6) | No Text (Arms 3+4+7+8) | Reminder (Arms 1+3+5+7) | No Reminder (Arms 2+4+6+8)
Number analyzed (Participants) | 2631 | 2613 | 2628 | 2616 | 2617 | 2627
Participants | 506 | 492 | 593 | 405 | 559 | 439

3. Secondary Outcome: Colorectal Cancer (CRC) Screening Completion (Any)
Description: Percent of patients who complete any CRC screening
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Box (Arms 1+2+3+4) | Envelope (Arms 5+6+7+8) | Text (Arms 1+2+5+6) | No Text (Arms 3+4+7+8) | Reminder (Arms 1+3+5+7) | No Reminder (Arms 2+4+6+8)
Number analyzed (Participants) | 2613 | 2631 | 2628 | 2616 | 2617 | 2627
Participants | 650 | 640 | 739 | 551 | 700 | 590

4. Secondary Outcome: FIT Positive Follow-up Scheduling
Description: Percent of patients with FIT+ results that schedule a colonoscopy
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Patients With a Positive FIT Result: Patients with a Positive FIT Result across all study arms.
Arm/Group | Patients With a Positive FIT Result
Number analyzed (Participants) | 50
Participants | 26

5. Secondary Outcome: FIT Positive Follow-up Completion
Description: Percent of patients with FIT+ results that complete a diagnostic colonoscopy
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With a Positive FIT Result
Number analyzed (Participants) | 50
Participants | 23

ADVERSE EVENTS:
Time Frame: Only All-Cause Mortality monitored/assessed up to 6 months from study start.
Description: Only All-Cause Mortality monitored/assessed up to 6 months from study start. The research solely tested methods of outreach for getting patients to complete mailed FIT for colorectal cancer screening. No drug, medical device, or medical procedure was under investigation.
Arm/Group | Arm 1: Box + Text + Reminder | Arm 2: Box + Text + No Reminder | Arm 3: Box + No Text + Reminder | Arm 4: Box + No Text + No Reminder | Arm 5: Standard Mail + Text + Reminder | Arm 6: Standard Mail + Text + No Reminder | Arm 7: Standard Mail + No Text + Reminder | Arm 8: Standard Mail + No Text + No Reminder
All-Cause Mortality (participants affected / at risk) | 0/656 | 0/661 | 0/653 | 0/661 | 1/655 | 0/656 | 0/653 | 1/649
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-11): https://cdn.clinicaltrials.gov/large-docs/22/NCT05341622/Prot_SAP_000.pdf